CLINICAL TRIAL: NCT02497040
Title: Effects of Scalp Block With Bupivacaine Versus Levobupivacaine on Haemodynamic Response to Head Pinning and Efficacy on Postoperative Analgesia
Brief Title: The Effects of Scalp Block With Bupivacaine Versus Levobupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, banu otlar can, anesthesia and reanimation, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: uludagu
Record Dates: First submitted 2015-07-02; First posted 2015-07-14 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
Keywords: anaesthesia; local anaesthesia; hemodynamics; bupivacaine; levobupivacaine
MeSH Terms: conditions — Hypertension | interventions — Levobupivacaine; Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- bupivacaine,levobupivacaine (Experimental): 20 ml of 0.5% bupivacaine 20 ml of 0.5% levobupivacaine
  Interventions: Drug: Levobupivacaine; Drug: Bupivacaine
- levobupivacaine (Active Comparator): 20 ml of 0.5% levobupivacaine saline as a placebo
  Interventions: Drug: Levobupivacaine; Drug: placebo
- bupivacaine (Active Comparator): 20 ml of 0.5% bupivacaine saline as a placebo
  Interventions: Drug: Bupivacaine; Drug: placebo

INTERVENTIONS:
Drug: Levobupivacaine — local injection
  Other Names: chirocaine
  Arms: bupivacaine,levobupivacaine; levobupivacaine
Drug: Bupivacaine — local injection
  Other Names: marcaine
  Arms: bupivacaine; bupivacaine,levobupivacaine
Drug: placebo — local injection
  Other Names: saline
  Arms: bupivacaine; levobupivacaine

SUMMARY:
Ninety American Society of Anesthesiologists (ASA) Physical Status classification system I-II patients were recruited for a randomised, placebo-controlled, double-blind study and were randomly divided into three groups to receive either 20 ml of 0.5% bupivacaine (Group B; n=30), 20 ml of 0.5% levobupivacaine (Group L; n=30) or saline as a placebo (Group C; n=30). Scalp block was performed 5 min before head pinning. The primary outcome of the study was mean arterial pressure (MAP) and secondary outcomes were heart rate (HR), visual analogue scale (VAS) scores, additional intraoperative and postoperative drug use. Postoperative pain was evaluated using a 10-cm visual analogue scale (VAS).

DETAILED DESCRIPTION:
Following approval from the Research Ethics Committee of the Medical Faculty of Uludağ University, (the date and protocol number assigned by this ethics committee were March 4, 2008 and 5/30, respectively),written informed consent was obtained from patients undergoing elective scheduled operations involving craniotomy during anaesthesia consultations. Ninety American Society of Anesthesiologists (ASA) Physical Status classification system I or II patients of either sex between 18-85 years of age were allocated to this randomised, prospective, placebo-controlled, double-blind study. The patients were randomly divided into three groups using a sealed-enveloped technique to receive either 20 ml of 0.5% bupivacaine (Group B (n=30)), 20 ml of 0.5% levobupivacaine (Group L (n=30)) or saline as a placebo (Group C (n=30)). Twenty-millilitre syringes for the block were prepared and numbered by a blinded assistant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status classification system 1-2

Exclusion Criteria:

* Uncontrolled hypertension, arrhythmia, diabetes mellitus or coagulopathy, coronary artery disease or a proven or suspected allergy to bupivacaine or levobupivacaine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: hulya bilgin, Study Director — uludag university anaesthesia and reanimation department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinosky ML, Fishman RL, Reeves ST, Harvey SC, Patel S, Palesch Y, Dorman BH. The effect of bupivacaine skull block on the hemodynamic response to craniotomy. Anesth Analg. 1996 Dec;83(6):1256-61. doi: 10.1097/00000539-199612000-00022. PMID 8942596
- [Background] Agarwal A, Sinha PK, Pandey CM, Gaur A, Pandey CK, Kaushik S. Effect of a subanesthetic dose of intravenous ketamine and/or local anesthetic infiltration on hemodynamic responses to skull-pin placement: a prospective, placebo-controlled, randomized, double-blind study. J Neurosurg Anesthesiol. 2001 Jul;13(3):189-94. doi: 10.1097/00008506-200107000-00002. PMID 11426091
- [Background] Costello TG, Cormack JR, Mather LE, LaFerlita B, Murphy MA, Harris K. Plasma levobupivacaine concentrations following scalp block in patients undergoing awake craniotomy. Br J Anaesth. 2005 Jun;94(6):848-51. doi: 10.1093/bja/aei135. Epub 2005 Apr 7. PMID 15817709

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine: 20 ml of 0.5% levobupivacaine saline as a placebo
  Bupivacaine: local injection
  placebo: local injection
Period: Overall Study
Arm/Group | Bupivacaine,Levobupivacaine | Levobupivacaine | Bupivacaine
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine,Levobupivacaine | Levobupivacaine | Bupivacaine | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 27 | 78
  >=65 years | 5 | 4 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 19 | 53
  Male | 15 | 11 | 11 | 37
Region of Enrollment [Number; unit: participants]
  Turkey | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Arterial Pressure
Time Frame: 220+-70 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bupivacaine,Levobupivacaine | Levobupivacaine | Bupivacaine
Number analyzed (Participants) | 30 | 30 | 30
mmHg | 110 (20) | 105 (20) | 100 (20)

ADVERSE EVENTS:
Arm/Group | Bupivacaine,Levobupivacaine | Levobupivacaine | Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine,Levobupivacaine (N=30) | Levobupivacaine (N=30) | Bupivacaine (N=30)
nause, vomitting,hypertensıon (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No